CLINICAL TRIAL: NCT01395589
Title: Rapid vs Maintenance Vitamin D Supplementation in Deficient Children With Asthma to Prevent Exacerbations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Khalid Ibrahim, Consultant, Hamad Medical Corporation
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1036
Record Dates: First submitted 2011-06-29; First posted 2011-07-15 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Asthma; Vitamin D Deficiency
Keywords: allergy; clinical trial; exacerbation; pediatrics
MeSH Terms: conditions — Asthma; Vitamin D Deficiency; Hypersensitivity | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Injectable + oral vitamin D (Active Comparator): Children with moderate-to-severe asthma exacerbations and vitamin D levels < 25 ng/mL.
  Interventions: Drug: Vitamin D
- Oral-only Vitamin D (Active Comparator): Children with moderate-to-severe asthma exacerbations and vitamin D levels < 25 ng/mL.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Children with moderate-to-severe asthma exacerbations and vitamin D levels < 25 ng/mL underwent masked randomization, and then open dosing to either IM+oral (the latter daily) therapy or daily oral-only therapy, and were followed for 12 months.

SUMMARY:
The role of vitamin D in respiratory health remains uncertain. Whether vitamin D reduces clinically important exacerbations of childhood asthma remains uncertain. We compared rapid to maintenance vitamin D repletion analyzed by baseline vitamin D level.

DETAILED DESCRIPTION:
Recently published Cochrane metaanalysis suggested that vitamin D reduces the risk of severe asthma exacerbations, but only 22 children contributed to that analysis from a study that found no difference in acute care visits or rescue steroid administration. Altogether, randomized trials performed in children show promise solely in meta-analyses that use varied clinical outcomes and analysis approaches.

Were vitamin D supplementation beneficial for children with asthma, it might prevent moderate to severe asthma exacerbations entirely in some children, reduce the overall frequency of exacerbations in a treated group, or both. To examine these possibilities, we designed a randomized explanatory study comparing rapid vs maintenance vitamin D supplementation for children with moderate-to-severe asthma and with low baseline vitamin D levels .

Children presenting to the ED with moderate-to-severe asthma exacerbations and vitamin D levels < 25 ng/mL underwent masked randomization, and then open dosing to either IM+oral (the latter daily) therapy or daily oral-only therapy, and were followed for 12 months.The primary outcome was patient-initiated unplanned visits for asthma exacerbations,examined two ways: cumulative proportions with an exacerbation, and average exacerbation frequency. As this was a nutrient study, we analyzed treatment groups by quartile of baseline vitamin D level, collecting repeat levels and clinical observations at 3, 6, 9,and 12 months after enrollment.

One hundred and sixteen patients in the IM+oral cohort vs 115 in the oral-only cohort had similar mean (SD) baseline levels: 15.1 (5.4) vs 15.8 (5.2) ng/mL (range, 3-25 ng/mL). There was no difference in the primary outcome over the entire 12-month observation period. However, rapid IM+oral supplementation significantly reduced unplanned visits for asthma exacerbations for children with baseline levels of 3 to 11 ng/mL during the initial 3 months: the relative exacerbation rate for the IM+oral cohort compared with the oral-only cohort at 3 months was 0.48 (95% CI, 0.28-0.89; P ¼ .008); average exacerbation frequency per child analysis, relative rate 0.36 (95% CI, 0.13-0.87; P ¼ .017).

So Rapid compared to maintenance vitamin D supplementation for children with the lowest levels resulted in short- but not long-term reduction in asthma exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Children 2-14 years of age with moderate to severe asthma and proved to be Vitamin D deficient by serum level.

EXCLUSION CRITERIA:

* Prematurity (Gestational age 34 weeks or less)
* Patients on vitamin D therapy
* Patients on seizure medication or diuretics
* Patients on chronic steroid use for other reasons than asthma
* Patient with chronic liver or kidney disease
* Patients with inherited bone disease
* Patients with hypo or hyper parathyroidism
* Patients with history of chronic lung disease other than asthma

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 597 (Actual)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Acute asthma exacerbations avoidable events . | 12 month
  Rapid compared to maintenance oral supplementation with vitamin D significantly reduced unplanned visits for asthma exacerbations for children with baseline levels of 3 to 11 ng/mL during the initial 3 months of treatment but not thereafter.

SECONDARY OUTCOMES:
Daily symptom burden differ in slow versus rapid vitamin D deficiency correction in patients with moderate to severe asthma | 12 month
  Rapid compared to maintenance vitamin D supplementation for children with the lowest levels resulted in short- but not long-term reduction in asthma exacerbations.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Khalid Al-Ansari, Study Chair — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Pediatric Emergency Center,Alsaad., Doha, Qatar